CLINICAL TRIAL: NCT06567600
Title: Combined Therapy Using Low-dose Gemcitabine and Cisplatin Chemotherapy and PD-1/PD-L1Antibody for Patients With Advanced and Unresectable Intrahepatic Cholangiocarcinoma: an Open-label, Multicenter, Single-arm Clinical Trial
Brief Title: Low-dose Gemcitabine and Cisplatin and PD-1/PD-L1 Antibody Therapy in Intrahepatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Linsen Ye, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSSY-2407
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Intrahepatic Cholangiocarcinoma; Chemotherapy Effect; Immunotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: low-dose gemcitabine and cisplatin combined with PD-1/PD-L1 inhibitors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose Gemcitabine and Cisplatin Chemotherapy plus PD-1/PD-L1Antibody (Experimental): Low-dose Gemcitabine and Cisplatin Chemotherapy:
  Gemcitabine 500 mg/m2 Cisplatin 12.5 mg/m2 on day 1 and day 8 of each 21-day cycle for up to eight cycles
  PD-1/PD-L1Antibody:
  Pembrolizumab 200mg on day 1 of each 21-day cycle Durvalumab 1500 mg on day 1 of each 21-day cycle After completion of gemcitabine and cisplatin, 200mg of Pembrolizumab or 1500 mg of Durvalumab may administer once every 3 or 4 weeks until clinical or imaging (per RECIST v1.1) disease progression or until unacceptable toxicity, withdrawal of consent, or any other discontinuation criteria were met.
  Interventions: Drug: Low-dose Gemcitabine and Cisplatin Chemotherapy plus PD-1/PD-L1Antibody

INTERVENTIONS:
Drug: Low-dose Gemcitabine and Cisplatin Chemotherapy plus PD-1/PD-L1Antibody — Low-dose Gemcitabine and Cisplatin Chemotherapy:
  Gemcitabine 500 mg/m2 Cisplatin 12.5 mg/m2 on day 1 and day 8 of each 21-day cycle for up to eight cycles
  PD-1/PD-L1Antibody:
  Pembrolizumab 200mg on day 1 of each 21-day cycle Durvalumab 1500 mg on day 1 of each 21-day cycle After completion of gemcitabine and cisplatin, 200mg of Pembrolizumab or 1500 mg of Durvalumab may administer once every 3 or 4 weeks until clinical or imaging (per RECIST v1.1) disease progression or until unacceptable toxicity, withdrawal of consent, or any other discontinuation criteria were met.
  Other Names: LDGC-PB

SUMMARY:
In this phase 2 study, researchers aimed to evaluate the efficacy and safety of low-dose gemcitabine and cisplatin chemotherapy and the immune checkpoint inhibitor PD-1/PD-L1 antibody in patients with advanced and unresectable intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
More and more studies suggest that low-dose chemotherapy has the ability to reshape the tumor microenvironment and promote tumor immunotherapy in a variety of tumors, supporting the rationality of combining low-dose chemotherapy with immunotherapy to effectively treat tumors with low T cell infiltration. More than half of intrahepatic cholangiocarcinomas are non-inflammatory "cold tumors", and their unique immunosuppressive microenvironment is one of the reasons for the poor response rate to immunotherapy. Low-dose chemotherapy can transform "cold" tumors with low immunogenicity and poor immune cell infiltration into "hot" tumors with immune responsiveness and sufficient immune cell infiltration, enhance the effect of ICIs on tumor cells, and minimize systemic toxicity, thus preserving a "therapeutic window" for combined immunotherapy/targeted therapy. Preclinical and clinical studies have shown that it is necessary to study the optimal dose of chemotherapeutic drugs in combination therapy. In combination therapy, long-term, adequate doses of chemotherapeutic drugs may be unnecessary because this will not only lead to more severe toxicity, but also damage rather than enhance anti-tumor immunity.

To determine the efficacy and safety of low-dose chemotherapy combined with PD-1/PD-L1 inhibitors in the treatment of patients with advanced intrahepatic cholangiocarcinoma, we designed an open-label, prospective, multicenter, single-arm clinical study of low-dose gemcitabine + cisplatin combined with PD-1/PD-L1 inhibitors in the treatment of patients with advanced intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female;
2. Histopathologically confirmed intrahepatic cholangiocarcinoma;
3. TNM Staging≥Stage II (American Joint Committee on Cancer Prognostic Groups)
4. Presence of at least one measurable lesion assessed using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST version 1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Child-Pugh score ≤ 7;
7. Adequate organ function (neutrophil count of ≥1.5×10^9 cells/L, hemoglobin concentrations of ≥90 g/L, platelet cell count of ≥100×10^9 cells/L, bilirubin ≤1.5×ULN, Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 5×ULN, serum creatinine ≤ 1.5 x ULN, Thyroid stimulating hormone (TSH) ≤ 1 x ULN;
8. The patient must be required to sign an informed consent form;

Exclusion Criteria:

1. Patients who have received previous treatment with interventional therapy, radiotherapy, ablation, chemotherapy, targeted therapy, immunotherapy (PD-1, PD-L1, CLTA-4 antibody, etc), or surgery within the last 2 months;
2. Patients with other malignant tumors within the last 5 years, except for cured non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid carcinoma;
3. Active tuberculosis infection. Patients with active tuberculosis infection within 1 year prior to enrollment; had a history of active tuberculosis infection more than 1 year before enrollment, did not receive formal anti-tuberculosis treatment or tuberculosis is still active;
4. Active infection requiring systemic therapy;
5. Human immunodeficiency virus (HIV) positive;
6. Have an active, known, or suspected autoimmune disease. Subjects who require only hormone replacement therapy for hypothyroidism and skin diseases that do not require systemic therapy may be enrolled;
7. Suffering from high blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
8. Abnormal blood coagulation (INR >1.5, or PT>ULN+4s, or APTT >1.5 x ULN), with a bleeding tendency or receiving thrombolytic or anticoagulant therapy;
9. Pregnant or lactating women;
10. Participated in other trials within the last 4 weeks;
11. Has a history of allergy to platinum;
12. Other factors that may influence the safety of the subject or the compliance of the test by the investigator. Serious illnesses (including mental illness), severe laboratory tests, or other family or social factors that require combined treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  ORR according to RECIST 1.1 using investigator assessment

SECONDARY OUTCOMES:
Incidence of adverse events | 12 months
  Rate of participants with treatment-related adverse events as assessed by CTCAE v4.0
Deepness of response (DpR) | 12 months
  DpR according to RECIST 1.1 using investigator assessment
Disease control rate (DCR) | 12 months
  DCR according to RECIST 1.1 using investigator assessment
Overall Survival (OS) | 36 months
  OS is defined as the time from date of combined theray start to the date of death from any cause or to the date of last follow-up if patients are alive
Progression-free Survival (PFS) | 36 months
  From the beginning date of combined therapy to the date of disease progression. PFS according to RECIST 1.1 using investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ye Linsen, Professor, Study Chair — The third affiliated hospital of SYSU
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China